CLINICAL TRIAL: NCT01856764
Title: A Phase 2a, 15-Day, Randomized, Parallel Group, Double-Blind, Multi-Centre, Vehicle Controlled Trial to Assess the Efficacy and Local Safety of a Cream Containing 0.5% Roflumilast - a Phosphodiesterase Type 4 Inhibitor (PDE4i) Dermal Formulation - on Atopic Dermatitis Patients With Skin Lesions of Moderate Severity
Brief Title: Topical Roflumilast in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROF-DERM_203; 2012-003000-12 (EudraCT Number); U1111-1133-6455 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5% Roflumilast Cream (Experimental): Roflumilast 0.5%, cream, topically, twice daily for up to 15 days.
  Interventions: Drug: 0.5% Roflumilast Cream
- Vehicle Cream (Placebo Comparator): Roflumilast formulation vehicle, cream, topically, twice daily for up to 15 days.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: 0.5% Roflumilast Cream — Roflumilast 0.5% cream
  Arms: 0.5% Roflumilast Cream
Drug: Vehicle Cream — Roflumilast formulation vehicle
  Arms: Vehicle Cream

SUMMARY:
The purpose of this study is to evaluate the effect of topical roflumilast on the reduction of atopic dermatitis lesions in adults with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female between 18 to 65 years of age, inclusive, with atopic dermatitis (AD) meeting Hanifin and Rajka's criteria.
2. Has lesional skin areas of moderate severity characterized by modified local SCORing Atopic Dermatitis (SCORAD) of at least 4, with an erythema score ≥2, and confirmed by a qualified investigator.
3. Has an index/target lesion of moderate severity approximately 20 cm^2, suitable for topical treatment.
4. Is willing to wash out from AD current active therapy prior to entry in the study.
5. Is willing and able to apply the study medication as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
6. If a male who is nonsterilized and sexually active with a female partner of childbearing potential, agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
7. If a female of childbearing potential who is sexually active with a nonsterilized male partner, agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
8. Is capable of understanding and complying with protocol requirements in the opinion of the investigator.
9. Signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. Has received any investigational compound within 30 days, or within 5 half-lives of the compound (whichever is longer) prior to the Screening visit.
2. Has a history of AD unresponsive or poorly responsive to topical treatments.
3. Has a history of hypersensitivity to phosphodiesterase (PDE)-4 inhibitors or to drugs of similar chemical classes or any inactive ingredients of the trial medication.
4. Has clinically significant abnormal hematological parameters of hemoglobin, hematocrit or erythrocytes at Screening, in the judgment of the investigator.
5. Has a history or current clinically relevant allergy or idiosyncrasy to drugs or food.
6. Had extensive exposure to ultraviolet (UV) light in the 4 weeks prior to first application of study medication, including tanning and sun beds or is intending to have such exposure during the study treatment that may interfere with the study assessments as judged by the investigator.
7. Has evidence of oozing of target lesion.
8. Has a current skin complication such as erythroderma or overt bacterial or viral infection for which treatment with anti-infectives are indicated.
9. Had systemic treatment with corticosteroids or retinoids for studied condition within 3 months prior to the first application of study medication.
10. Had topical or transdermal treatments, such as but not limited to retinoids, nicotine or hormone replacement therapies, on or near the intended site of application within 4 weeks prior to first application of study medication.
11. Had treatment with systemic/locally acting medications/procedures that might counter or influence the study aim within 4 weeks prior to first application of study medication and during the study (e.g., anti-histamines).
12. Has used emollients/moisturizers on areas to be treated within 24 hours prior to the first application of study medication.
13. Has used biologics at any time for treatment of AD.
14. Is currently enrolled in an investigational drug or device study.
15. Has any clinically significant illness that may influence the outcome of the trial from 4 weeks before Day 1 through trial completion.
16. Has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) values greater than 2.0 × upper limit of normal (ULN), or other clinically significant abnormal laboratory test that, in the opinion of the Investigator, would compromise the participant's ability to safely complete the trial.
17. Has a significant medical condition and/or conditions that, in the opinion of the Investigator, would interfere with the treatment, safety or compliance with the protocol.
18. Has a history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
19. Has a history of alcoholism or illicit drug abuse within 5 years prior to the Screening Visit or is currently consuming >14 alcoholic drinks per week.
20. If female, is pregnant, nursing or planning a pregnancy during the study period.
21. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study medication. This criterion does not apply to those participants with successfully resected basal cell or stage I squamous cell carcinoma of the skin.
22. Has a chronic or clinically relevant acute infection.
23. Has a history of depression associated with suicidal ideation and behavior.
24. Has hemodynamically significant cardiac arrhythmias or heart valve deformations.
25. Is an immediate family member, a study site employee, in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or at risk for consenting under duress.
26. Was institutionalized because of a legal or regulatory order.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (3):
- Germany (3):
  - Berlin
  - Gera
  - Hamburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 centers in Germany from 10 June 2013 to 18 March 2014.
Pre-assignment Details: Participants with a historical diagnosis of Atopic Dermatitis were enrolled in 1 of 2 twice daily (BID) treatment groups.
Period: Overall Study
Arm/Group | 0.5% Roflumilast Cream | Vehicle Cream
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% Roflumilast Cream | Vehicle Cream | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (11.50) | 36.5 (9.65) | 34.6 (10.66)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Germany | 20 | 20 | 40
Height [Mean (Standard Deviation); unit: centimeters] | 177.3 (9.27) | 174.9 (10.13) | 176.1 (9.66)
Weight [Mean (Standard Deviation); unit: kilograms] | 81.72 (21.757) | 78.31 (12.965) | 80.02 (17.762)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.65 (5.007) | 25.59 (3.477) | 25.62 (4.255)
Smoking Classificaiton [Number; unit: participants]
  Never smoked | 5 | 8 | 13
  Current smoker | 10 | 9 | 19
  Ex-Smoker | 5 | 3 | 8
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 0 | 0 | 0
  Surgically sterile | 0 | 0 | 0
  Female of childbearing potential | 9 | 11 | 20
  N/A (male participant) | 11 | 9 | 20
Baseline Modified Local SCORing Atopic Dermatitis (SCORAD) [Mean (Full Range); unit: scores on a scale] | 5.60 [4.0 to 8.0] | 5.85 [4.0 to 8.0] | 5.725 [4.0 to 8.0]
Baseline Transepidermal Water Loss (TEWL) Mean [Mean (Full Range); unit: g/m^2/hr] | 41.47 [17.8 to 69.8] | 41.57 [17.8 to 63.3] | 41.52 [17.8 to 69.8]
Baseline Participant Assessment of Pruritis [Mean (Full Range); unit: scores on a scale] | 5.05 [0.0 to 9.0] | 5.00 [2.0 to 10.0] | 5.025 [0.0 to 10.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 15 in Modified Local SCORing Atopic Dermatitis (SCORAD)
Description: Modified Local SCORAD is the sum of 5 individual indexes; erythema, edema/papulation, oozing/crusts, excoriations and lichenification scored on a 4 point scale, where 0=absent and 3=severe, with a total possible score of 15. Higher scores indicate greater severity.
Time Frame: Baseline and Day 15
Population: All randomized participants who received at least one application of any double-blind study medication with a score at Day 15. One subject in the 0.5% Roflumilast group was missing Day 15 data.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 0.5% Roflumilast Cream | Vehicle Cream
Number analyzed (Participants) | 19 | 20
Scores on a scale | -2.30 (0.354) | -1.75 (0.347)
Statistical Analysis 1: Comparison: 0.5% Roflumilast Cream vs Vehicle Cream; Test type: Superiority or Other; p = 0.276, Mixed Models Analysis — Mixed Model Repeated Measures (MMRM) Model: SCORAD change from baseline = treatment + visit + treatment by visit interaction + baseline SCORAD score; LS Mean Difference = -0.55, 95% CI 2-sided [-1.5542 to 0.4574], Standard Error of Mean 0.496

2. Secondary Outcome: Change From Baseline to Day 15 in Transepidermal Water Loss (TEWL) Values
Description: Diffusion of water through the skin is measured using a Tewameter. At each visit, 3 measurements are taken per treatment area (at 3 different areas of the target lesion). The TEWL value at each visit is the average of these measurements.
Time Frame: Baseline and Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/m^2/hr
Arm/Group | 0.5% Roflumilast Cream | Vehicle Cream
Number analyzed (Participants) | 19 | 20
g/m^2/hr | -18.60 (2.467) | -12.69 (2.417)
Statistical Analysis 1: Comparison: 0.5% Roflumilast Cream vs Vehicle Cream; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis — MMRM model: TEWL change from baseline = treatment + visit + treatment by visit interaction + baseline TEWL score; LS Mean Difference = -5.91, 95% CI 2-sided [-12.9134 to 1.0835], Standard Error of Mean 3.454

3. Secondary Outcome: Change From Baseline to Day 15 in Participants' Assessment of Pruritus
Description: Severity of pruritus is assessed by the participants and recorded on a numeric scale ranging from 0 to 10, where 0 indicates the absence of the symptoms and 10 indicates the most severe symptoms.
Time Frame: Baseline and Day 15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 0.5% Roflumilast Cream | Vehicle Cream
Number analyzed (Participants) | 19 | 20
Scores on a scale | -3.05 (0.426) | -1.50 (0.417)
Statistical Analysis 1: Comparison: 0.5% Roflumilast Cream vs Vehicle Cream; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — MMRM model: Assessment of Pruritus change from baseline = treatment + visit + treatment by visit interaction + baseline Assessment of Pruritus score; LS Mean Difference = -1.56, 95% CI 2-sided [-2.7656 to -0.3492], Standard Error of Mean 0.596

ADVERSE EVENTS:
Time Frame: From the time informed consent is signed through 7 days after the last dose of study drug (up to Day 22)
Description: The population consisted of all randomized participants. At each visit, investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment
Arm/Group | 0.5% Roflumilast Cream | Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5% Roflumilast Cream (N=20) | Vehicle Cream (N=20)
Application Site Pain (General disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Red blood cells urine (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.